CLINICAL TRIAL: NCT00243126
Title: Family-based HIV Prevention for Adolescent Females
Brief Title: Family-based HIV Prevention for Adolescent Girls
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); National Institute of Mental Health (NIMH) (NIH); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: ATN 012
Record Dates: First submitted 2005-10-19; First posted 2005-10-21 (Estimated); Last update posted 2017-03-01 (Actual); Status verified 2016-02

CONDITIONS: HIV Infections
Keywords: HIV prevention; HIV Seronegativity; HIV negative
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Family-Based Risk Reduction Intervention (Experimental): The intervention will be delivered in five, two-hour, small group sessions, across five weeks (group will meet once per week). Each of the 5 modules consists of 3 sessions: a one-hour session for the daughters meeting together with each other, a one-hour session for the mothers meeting together with each other; and a one-hour session in which the daughters and mothers meet together. Therefore, each week, the daughters will meet as a group for one hour of each module, while the mothers meet as a group for one hour, and for one hour the mothers and daughters will all meet together.
  Interventions: Behavioral: Family-Based Risk Reduction Intervention
- No Treatment Control Group Condition (No Intervention): A no treatment control group condition will be utilized for this preliminary feasibility study. Participants in this condition, both mothers and adolescents will be assessed at baseline, immediate post-intervention, at 3-month follow-up and at 6-month follow-up.

INTERVENTIONS:
Behavioral: Family-Based Risk Reduction Intervention — The intervention module topics include five modules and each module is 2 hours in length. The intervention will focus on the elements critical to HIV risk behavior change. These include: risk education (practical understanding of factors responsible for risk and behavior changes needed to reduce risk); threat personalization (accurate appraisal of personal risk based on behavior); self-efficacy (belief that one can implement risk reduction behavior changes and that if changes are made they will have protective value); skills acquisition (e.g., condom use, safer sex guidance, negotiation); cognitive problem-solving skills; and reinforcement.
  Arms: Family-Based Risk Reduction Intervention

SUMMARY:
This is an exploratory/developmental study to support the early phases of development and evaluation of a family-based HIV prevention program for adolescent girls prior to a full-scale trial. Research on the new intervention will include evaluating the feasibility, tolerability, and acceptability of the intervention, and allow us to obtain the preliminary data needed as a pre-requisite to a larger-scale intervention study.

Adolescent females and their mother/guardian will be randomized to either: a family-based risk reduction intervention; or a no-treatment control group condition. Participants in both conditions will be assessed at baseline, immediate post-intervention, and at 3- and 6-month follow-ups. A subset of families (12 adolescents and 12 mothers) will participate in a qualitative interview following the 6-month follow-up, in which information will be obtained on participant perception of procedures and intervention content, and whether they have utilized skills taught following the end of the project.

DETAILED DESCRIPTION:
Participants will be involved with the study and follow up for a total of 32 to 36 weeks.

68-84 female adolescents and their mother/guardian (total N = 136-168).

African American or mixed race, sexually active female adolescents age 15 to 19 who are at risk for HIV infection and their mother/guardian

The adolescent participant and her mother/guardian will be randomized to either a family-based risk reduction intervention or a no-treatment control group condition.

Participants in both conditions will be assessed at baseline, immediate post-intervention, and at 3- and 6-month follow-ups. A subset of 24 participants from the intervention condition (12 adolescents and 12 mothers) will participate in a qualitative interview following the 6-month follow-up, in which information will be obtained on participant perception of procedures and intervention content, and whether they have utilized skills taught following the end of the project.

Interviewers will collect participant data from the baseline and follow-up behavioral interviews using a Computer Assisted Personal Interviewing (CAPI) method on a portable computer.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Between the age of 15 years and 0 days and 19 years and 364 days at the time of initial eligibility screening.
* Born in the United States
* Self identifies as all or part African American.
* Sexually active, defined as having had vaginal or anal intercourse
* Has engaged in unprotected sex during the past 3 months
* Is willing to invite and participate with her mother/guardian in the intervention
* Has either a biological mother or a guardian who is willing to participate in the study and meets the eligibility criteria

For the purposes of this pilot study, biological mothers are eligible, as are non-biological primary caretakers serving as mother/guardians who have guardianship of the adolescent and with whom the adolescent is living.

* Able to understand spoken and written English sufficiently to provide assent/consent and to be interviewed and participate in the study intervention.
* Not intending to relocate out of the current geographical area for the duration of study participation.
* Provides informed assent or consent

Mother or Mother/guardian

* Has legal guardianship; and
* Currently resides with the adolescent.
* Self identifies as all or part African American.
* Born in the United States
* Able to understand spoken and written English sufficiently to provide consent and to be interviewed and participate in the study intervention.
* Not intending to relocate out of the current geographical area for the duration of study participation.
* Provides informed consent

Exclusion Criteria:

* Adolescent is currently pregnant or has carried a pregnancy to term
* Adolescent self-reports as HIV positive

Ages: 15 Years to 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 168 (Actual)
Dates: Start 2005-11; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Test the feasibility of implementing intervention | 32-26 Weeks
  The primary objective of this pilot study is to test the feasibility of implementing a mother-daughter HIV risk reduction intervention for at-risk female adolescents.

SECONDARY OUTCOMES:
Conduct a preliminary efficacy test of the intervention | 32-36 Weeks
  The secondary objective of this pilot study is to conduct a preliminary efficacy test of the intervention to determine if trends towards significant effects for reducing unprotected sex and/or reducing substance use are found.

CONTACTS AND LOCATIONS:
Overall Officials: Debra A Murphy, Ph.D., Study Chair — University of California, Los Angeles
Locations (2):
- United States (2):
  - John H. Stroger Jr. Hospital and the Core Center, Chicago, Illinois
  - Mount Sinai Adolescent Health Center, New York, New York

REFERENCES:
- See also: Website for the Adolescent Trials Network for HIV/AIDS Interventions — http://www.atnonline.org